CLINICAL TRIAL: NCT01846949
Title: Study for Clinical Significance of Use of Alphafetoprotein (AFP), AFP-L3 and Des-gamma-carboxy Prothrombin (DCP) Versus US Alone in Surveillance for HCC
Brief Title: Surveillance Study for HCC by Combining Biomarkers With Imaging (ALDUS)
Acronym: ALDUS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: ALDUS Study Group (Other)
Responsible Party: Sponsor
Other Study IDs: ALDUS
Record Dates: First submitted 2013-04-23; First posted 2013-05-06 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is intended to be a prospective observational study at multiple sites, not a randomized controlled trial (RCT). The uses of the biomarkers has been approved by government regulations and adopted for surveillance programs in some countries, thus an RCT which compares patients followed by US alone with patients followed by both US and the biomarkers would raise an ethical conflict, especially in countries where the biomarkers have been routinely used.

For this study, enrolled patients will be followed by US and the biomarkers at regular intervals and classified after completing the study to evaluate the clinical effectiveness of the biomarkers. The comparisons of sensitivity, specificity, and other parameters with respect to tumor characteristics will be made among US alone, the biomarkers, and combined use of US and the biomarkers. Also economical effectiveness of using the biomarkers will be investigated in this study.

Requirement status is monitored every month.

DETAILED DESCRIPTION:
Data are being stored in the electric data capture (EDC) server.

ELIGIBILITY:
Inclusion Criteria:

* Patients with compensated cirrhosis. No discrimination by underlying causes will done.
* Patients aged 18 years and older
* Patients agree to the informed consent

Exclusion Criteria:

* Patients with liver cancer at the time of enrollment
* Patients who have experienced HCC or other malignant tumor with in five (5) years
* Women with pregnancies
* Patients who are likely to be transplanted within one (1) year
* Patients with ≥ 3 mg/dL of total bilirubin
* Patients with uncontrollable ascites
* Patients with ≥ Grade II of hepatic encephalopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with compensated cirrhosis.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-05; Primary Completion 2021-12 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Hepatocellular carcinoma | Expected time frame; 2.5 years
  Tumor marker measurement and ultrasonography are conducted at an interval of 13 weeks, until total events (HCC occurrence) reach to 120 cases.

SECONDARY OUTCOMES:
Survival | 2 and 5 year after patient enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Graduate School of Medicine and Faculty of Medicine, The University of Tokyo, Tokyo, Japan